CLINICAL TRIAL: NCT00636441
Title: A Randomized Phase II Trial Evaluating the Performance of Genomic Expression Profiles to Direct the Use of Preoperative Chemotherapy for Early Stage Breast Cancer
Brief Title: Trial to Evaluate Genomic Expression Profiles to Direct Preoperative Chemotherapy in Early Stage Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to reproducibility issues with genomics prediction model
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00001345; W81XWH-07-1-0394; BC060228-W81XWH-07-1-0394
Record Dates: First submitted 2008-03-09; First posted 2008-03-14 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2014-10

CONDITIONS: Early-Stage Breast Cancer
Keywords: Early-Stage Breast Cancer; Preoperative systemic chemotherapy (PST); Genomic; Genomic Predictor; Genomic Expression Profiles; Randomized; Pathologic complete response (pCR); HER2 negative; Doxorubicin and docetaxel; Doxorubicin and cyclophosphamide
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response | interventions — Doxorubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guided Arm (Active Comparator): Genomically-guided treatment allocation.
  This arm has the following cohorts:
  * AC sensitive patients [>60% probability of response to AC]
  * TC sensitive patients [>60% probability of response to TC]
  * Patients sensitive to neither AC nor TC; randomized to AC or TC
  Interventions: Drug: Doxorubicin/Cyclophosphamide (AC) or Docetaxel/Cyclophosphamide (TC)
- Non-Guided Arm (Active Comparator): Non-genomically-guided treatment allocation.
  This arm has the following cohorts:
  * In patients randomly assigned to AC:
    * Patients sensitive to AC
    * Patients sensitive to TC
    * Patients sensitive to neither AC nor TC
  * In patients randomly assigned to TC:
    * Patients sensitive to AC
    * Patients sensitive to TC
    * Patients sensitive to neither AC nor TC
  Interventions: Drug: Doxorubicin/Cyclophosphamide (AC) or Docetaxel/Cyclophosphamide (TC)

INTERVENTIONS:
Drug: Doxorubicin/Cyclophosphamide (AC) or Docetaxel/Cyclophosphamide (TC) — Doxorubicin 60 mg/m² and Cyclophosphamide 600 mg/m² (AC) or Docetaxel 75 mg/m² and Cyclophosphamide 600 mg/m² (TC) every 3 weeks for 4 cycles as neoadjuvant therapy
  Other Names: Adriamycin (Doxorubicin); Rubex (Doxorubicin); Taxotere (Docetaxel); Cytoxan (Cyclophosphamide)

SUMMARY:
This multi-center randomized Phase II study assigned HER2-negative early-stage breast cancer patients to receive preoperative systemic chemotherapy in either a "genomic-guided" arm or a "non-guided arm." The "genomic-guided" method (Arm 1) used genomic expression profiling to assign the preoperative therapy (Doxorubicin/Cyclophosphamide (AC) versus Docetaxel/Cyclophosphamide (TC), while Arm 2 used random assignment to these two therapies.

DETAILED DESCRIPTION:
Primary Objective 1 was to test for an arm difference in pathological complete response rates. Secondary Objective 2 was to estimate and test the difference in pathologic complete response rates between drug-sensitive patients who received their preferred drug and drug-resistant patients randomized to AC or TC.

Secondary objectives included: to determine the 60% cutoff for the genomic profiles resulted in a larger pathologic CR rate for the guided arm than for the unguided arm; to compare the pathologic CR rates of patients whose genomic predictive probabilities indicated that they were resistant to both chemotherapy regimens with the pathologic CR rates of patients whose genomic predictive probabilities indicated that they were sensitive to only one treatment and who were then randomly assigned to a treatment for which they were resistant (combining AC and TC subgroups); Secondary Objective 3 in patients with T2 and T3 tumors classified as requiring mastectomy at baseline, compare the guided and non-guided treatment arms on rates of breast conserving surgery with negative final margins; Secondary Objective in patients with T2 tumors classified as potential candidates for breast conservation, compare the guided and non-guided arms on rates of breast conserving surgery at first attempt; Secondary Objectives 5, 6, 7 and 8 to correlate genomic profiles (i.e., genomic predictive probabilities) with clinical response, disease-free survival, sites of recurrence, and overall survival; Secondary Objective 9:to compare the mean cost of guided versus non-guided treatment; and Secondary Objective 10 to assess patient perceptions of participating in a clinical trial that evaluated cancer genomics for preoperative systemic therapy of early-stage breast cancer.

Objective 10 details: Due to space limitations in the Outcome Measure Description field, details are supplied here:

To assess patient motivation and participation for study participation in a clinical trial evaluating cancer genomics for treatment patients provided responses for the following questions at both baseline (the day of chemotherapy start) and following post-surgical medical oncology evaluation:

One of the goals of this study is to tailor your cancer treatments for you based upon a genomic analysis of your tumor. How much did the knowledge that the treatment is potentially tailored specifically for your tumor influence your decision to participate in this study? (Select One)

Response 1: I did not know that the treatment was tailored.

Response 2: I do not understand what "tailored treatment based upon genomic analysis of "my tumor" means.

Response 3: The information that this was a tailored treatment based upon genomic analysis of my tumor decreased my willingness to participate in this study.

Response 4: The information that this was a tailored treatment based upon genomic analysis of my tumor was of neutral value in the decision making process to participate in this study and did not influence my decision to participate.

Response 5: The information that this was a tailored treatment based upon genomic analysis of my tumor played a minor role in helping me decide to participate in the study.

Response 6: The information that this was a tailored treatment based upon genomic analysis of my tumor played a major role in helping me decide to participate in the study.

Response 7: The information that this was a tailored treatment based upon genomic analysis of my tumor was the primary reason that I decided to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic Documentation: Patients must have a histologic (i.e., not just cytologic) diagnosis of invasive breast cancer by core biopsy. Excisional biopsy or incisional biopsy is not allowed. All breast cancer histologic types are allowed.
2. Stage: Any patient with a clinical T1c (>1.5 cm) to T3 invasive breast cancer by the revised TNM staging system (AJCC 6th edition) will be eligible. Any N stage disease is allowed. No distant metastases allowed.
3. Tumor Site: Patients must have invasive cancer in the breast. Multifocal disease (i.e. confined to a single quadrant in the same breast) is allowed. Multicentric disease (i.e. disease in multiple breast quadrants) is not allowed. Determination of multifocal and multicentric disease status will be made by the evaluating surgeon; ambiguous cases will be reviewed by the principal investigator. Patients with synchronous contralateral invasive breast cancers are not eligible; prior contralateral breast cancer allowed as long as patient has not received prior chemotherapy or radiation therapy in the past 5 years.
4. Measurable Disease: Patients must have measurable disease in the breast by imaging studies (mammogram, ultrasound, or MRI), and must be greater than 1.5 cm in at least one dimension by one or more of the imaging assessments.
5. Conventional Biomarker Status: Standard clinical biomarkers for ER, PR, and HER2 must be obtained on the initial diagnostic core biopsy. The invasive cancer must be HER2 negative (i.e. immunohistochemistry score 1-2+ and/or FISH non-amplified). Any ER/PR status is allowed. Patients who are HER2 2+ on initial immunohistochemistry assessment will be further assessed by FISH. In this instance, patient will be consented and further screened for eligibility and have tissue acquired for genomic profiling. If the standard of care additional FISH testing is positive for HER2 gene amplification, the patient will not be randomized and will be treated in the same manner as screen failures.
6. Must be deemed a surgical candidate.
7. Fresh tissue biopsy material must be available for genomics analysis.
8. No prior chemotherapy, radiotherapy, or biologic/targeted therapy for the currently diagnosed breast cancer, or any other malignancy in the past 5 years, is allowed. No prior anthracycline or taxane therapy.
9. Prior malignancies are allowed if the patient is considered to be disease-free for 5 or more years and is deemed to be at low risk for recurrence. Patients with any prior diagnosis of in situ malignancies (melanoma, bladder, colon, cervical, basal cell, or squamous carcinoma) are eligible regardless of time from diagnosis.
10. Aged at least 18 years.
11. ECOG Performance Status 0-1.
12. Adequate Organ Function:

    1. Total bilirubin ≤1.0 x the institutional ULN
    2. Hepatic enzymes (AST (SGOT), ALT (SGPT)) ≤1.5x the institutional ULN
    3. Alkaline Phosphatase ≤2.5 x ULN
    4. Serum creatinine ≤2.0 mg/dl
    5. Neutrophil count (ANC or AGC) ≥1000/ μL
    6. Platelets ≥100,000/ μL
    7. Cardiac Ejection Fraction ≥50% by MUGA, Echo or MRI.
13. Significant cardiac disease that would preclude the use of anthracyclines: No myocardial infarction in the last 6 months; history of congestive heart failure, serious cardiac arrhythmia requiring medication, active coronary artery disease/angina pectoris requiring therapy, uncontrolled hypertension defined as BP >150/90 despite medication; any other unstable cardiac condition as perceived by treating physician or study PI.
14. No other serious medical or psychiatric illness.
15. Pregnancy: Patients may not be pregnant or nursing at the time of enrollment and other restrictions apply.
16. Signed written informed consent including HIPAA.

Exclusion Criteria:

1. Patients who have received investigational drugs within 4 weeks prior to starting study drug and/or who have not recovered from side effects of such therapy are not eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul K Marcom, MD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Potti A, Dressman HK, Bild A, Riedel RF, Chan G, Sayer R, Cragun J, Cottrill H, Kelley MJ, Petersen R, Harpole D, Marks J, Berchuck A, Ginsburg GS, Febbo P, Lancaster J, Nevins JR. Genomic signatures to guide the use of chemotherapeutics. Nat Med. 2006 Nov;12(11):1294-300. doi: 10.1038/nm1491. Epub 2006 Oct 22. PMID 17057710 (Retraction: PMID 21217686 Potti A, Dressman HK, Bild A, Riedel RF, Chan G, Sayer R, Cragun J, Cottrill H, Kelley MJ, Petersen R, Harpole D, Marks J, Berchuck A, Ginsburg GS, Febbo P, Lancaster J, Nevins JR. Nat Med. 2011 Jan;17(1):135)

RESULTS

PARTICIPANT FLOW:
Groups:
- Guided AC Sensitive: Genomically-guided >60% probability of response to AC
  AC: Doxorubicin 60 mg/m² and Cyclophosphamide 600 mg/m² (AC) every 3 weeks for 4 cycles as neoadjuvant therapy
- Guided TC Sensitive: Genomically-guided treatment >60% probability of response to TC
  TC: Docetaxel 75 mg/m² and Cyclophosphamide 600 mg/m² (TC) every 3 weeks for 4 cycles as neoadjuvant therapy
- Guided AC Non-sensitive: Genomics guided treatment <60% probability of response to both AC and TC; randomized to AC
  AC: Doxorubicin 60 mg/m² and Cyclophosphamide 600 mg/m² (AC) every 3 weeks for 4 cycles as neoadjuvant therapy
- Guided TC Non-Sensitive: Genomics guided treatment <60% probability of response to both AC and TC; randomized to TC
  TC: Docetaxel 75 mg/m² and Cyclophosphamide 600 mg/m² (TC) every 3 weeks for 4 cycles as neoadjuvant therapy
- Non-guided AC: Non-genomics guided treatment; randomized to AC
  AC: Doxorubicin 60 mg/m² and Cyclophosphamide 600 mg/m² (AC) every 3 weeks for 4 cycles as neoadjuvant therapy
- Non-guided TC: Non-genomics guided treatment; randomized to TC
  TC: Docetaxel 75 mg/m² and Cyclophosphamide 600 mg/m² (TC) every 3 weeks for 4 cycles as neoadjuvant therapy
Period: Overall Study
Arm/Group | Guided AC Sensitive | Guided TC Sensitive | Guided AC Non-sensitive | Guided TC Non-Sensitive | Non-guided AC | Non-guided TC | Screen Failure
Started | 6 | 7 | 6 | 6 | 6 | 7 | 18
Assigned Treatment | 6 | 7 | 6 | 6 | 6 | 7 | 1 (This is a late determined ineligibility.)
Completed | 6 | 6 | 5 | 6 | 6 | 6 | 0
Not Completed | 0 | 1 | 1 | 0 | 0 | 1 | 18
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Late, ineligible | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 0 | 0 | 17

BASELINE CHARACTERISTICS:
Population: All patients who signed a consent form are included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Guided AC Sensitive | Guided TC Sensitive | Guided AC Non-sensitive | Guided TC Non-Sensitive | Non-guided AC | Non-guided TC | Screen Failure | Total
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 7 | 18 | 56
Age, Continuous [Median (Standard Deviation); unit: years] | 48.6 (8.7) | 51.2 (7.3) | 52.6 (8.0) | 48.8 (9.1) | 53.5 (6.7) | 58.9 (12.9) | 52.5 (13.0) | 52.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 6 | 6 | 6 | 7 | 18 | 56
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 6 | 6 | 6 | 7 | 18 | 56

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) Rate in Patients With HER2-negative Early-stage Breast Cancer
Description: Pathological complete response (pCR) was defined as the disappearance of all invasive disease in the breast or if only residual in situ or lymph node disease is found. The pCR rate is presented with its 95% confidence interval for the Guided and Non-guided arms.
Time Frame: 4-5 weeks after the fourth cycle of chemotherapy; approximately 16-17 weeks
Population: All eligible treated patients. The three patients not included are two who had allergic reactions to the assigned treatment, and one with metastatic disease on biopsy of a spine lesion at the end of assigned treatment so never went to surgery.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Guided Arm: Genomically-guided treatment allocation.
- Non-Guided Arm: Non-genomically-guided treatment allocation.
Arm/Group | Guided Arm | Non-Guided Arm
Number analyzed (Participants) | 24 | 11
percentage of participants | 16.7 [4.7 to 37.4] | 9.1 [0.2 to 41.3]

2. Secondary Outcome: Probabilities of Being Sensitive to AC and TC as Determined by the Patient's Genomic Signatures
Description: To determine in early stage breast cancer treated with PST whether genomic profiling can identify drug-sensitive and drug-resistant patients including a comparison of subgroups for the two individual regimens (i.e. AC and TC). To determine if the 60% cutoff for the genomic profiles is optimal in predicting the response to chemotherapy regimens.To describe the performance of the genomic profiles in assessing the relative responsiveness of: 1) Patients predicted to be resistant to both chemotherapy regimens; and 2) Patients randomly assigned to one treatment whose genomic profiles suggest receiving the other regimen (in both AC and TC subgroups).
Time Frame: 10 years
Population: This outcome is not summarized due to irreproducibility of the genomics-based prediction model and resulting probability estimates
Arm/Group | Guided Arm | Non-Guided Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Patients Who Had Breast-conserving Surgery With Negative Margins
Description: The percentage of patients who had breast-conserving surgery with negative margins, measured in patients with T2 and T3 tumors classified as requiring mastectomy at baseline.
Time Frame: 6 months
Population: Since final margin status was not collected, this analysis could not be done.
Arm/Group | Guided Arm | Non-Guided Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Percentage of Patients Who Had Breast-conserving Surgery at First Attempt.
Description: The percentage of patients who had breast-conserving surgery at first attempt, measured only in patients with T2 tumors classified as potential candidates for breast conservation.
Time Frame: 6 months
Population: Data from all eligible patients with non-missing values on this outcome were used.
Measure: Number (95% Confidence Interval); unit: percentage of T2 tumor patients
Arm/Group | Guided Arm | Non-Guided Arm
Number analyzed (Participants) | 3 | 1
percentage of T2 tumor patients | 67 [9 to 99] | 100 [NA to NA] — can not calculate confidence interval N of 1.

5. Secondary Outcome: Clinical Response Using WHO Criteria
Description: WHO criteria are based on the sum of the products of the longest axis and the longest perpendicular axis. Bi-dimensional measurements were taken of all breast lesions and axillary nodes using the best imaging modality performed after completion of assigned therapy.
  Clinical Complete Response (cCR): Disappearance of all target lesions by physical exam and best imaging modality.
  Clinical Partial Response (cPR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the sum LD at treatment initiation. Patients having a documented response with no reconfirmation of the response will be listed with stable disease.
  Progression (PD): At least a 20% increase in the sum of the LD of target lesions or the appearance of one or more new lesion.
Time Frame: 12 weeks, 2-3 weeks after the fourth cycle of chemotherapy
Population: All eligible treated patients were used in this analysis.
Measure: Number; unit: participants
Arm/Group | Guided Arm | Non-Guided Arm
Number analyzed (Participants) | 25 | 13
participants
  Complete Response (cCR) | 2 | 2
  Partial Response (cPR) | 15 | 7
  Stable Disease | 6 | 2
  Progressive Disease | 1 | 0
  Not Evaluable/Not Assessed | 1 | 2

6. Secondary Outcome: Disease-free Survival
Description: Disease-free survival is defined as the length of time from enrollment to local or distant disease recurrence, whichever comes first; disease-free deaths are censored. The 2-year disease-free survival rate is estimated with its 95% confidence interval.
Time Frame: 2 years
Population: All eligible treated patients were used in this analysis.
Measure: Number (95% Confidence Interval); unit: estimated % of participants disease-free
Arm/Group | Guided Arm | Non-Guided Arm
Number analyzed (Participants) | 25 | 13
estimated % of participants disease-free | 92 [71 to 98] | 89 [43 to 98]

7. Secondary Outcome: Sites of Recurrence
Description: Sites of Recurrence is a categorical outcome whose possible values are the organ-specific sites at which disease recurrence was observed. A patient may recur at more than one site.
Time Frame: 10 years
Population: All eligible treated patients. Four of these 38 participants experienced recurrence of their breast cancer; two of the four patients had multiple sites of recurrence.
Measure: Number; unit: participants
Arm/Group | Guided Arm | Non-Guided Arm
Number analyzed (Participants) | 25 | 13
participants
  Bone | 3 | 1
  Brain | 1 | 0
  Chest Wall | 1 | 0
  Liver | 2 | 0
  Lung | 1 | 0

8. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from enrollment to death due to any cause. The 2-year overall survival rate is estimated with the Kaplan-Meier method.
Time Frame: 2 years
Population: All eligible treated patients with known follow-up status.
Measure: Number (95% Confidence Interval); unit: Estimated % of participants surviving
Arm/Group | Guided Arm | Non-Guided Arm
Number analyzed (Participants) | 24 | 12
Estimated % of participants surviving | 96 [74 to 99] | 100 [NA to NA] — Since no deaths occurred on or before the 2-year time point a confidence interval cannot be estimated.

9. Secondary Outcome: Economic Impact of Using Genomic Assessment to Guide Management.
Description: Economic Impact (i.e., cost of care) will be calculated by first assessing the quantity of clinical resources used by each patient in the study arm, and then assigning a cost to each resource using cost information derived from a costing study to be undertaken outside of this protocol.
Time Frame: 5 years
Population: Since these data were not collected, this analysis could not be done.
Arm/Group | Guided Arm | Non-Guided Arm
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Patients' Perceptions of Participating in a Clinical Trial Evaluating Cancer Genomics for PST of Early-stage Breast Cancer.
Description: A short questionnaire was administered at baseline (the day chemotherapy was started) and following post-surgical medical oncology evaluation to assess the patient's understanding of the study being conducted, and the patient's expectations of the treatment. Due to space limitations, the full survey is presented in the Detailed Description.
Time Frame: 1 year
Population: The overall enrollment was insufficient to provide for any substantive analysis.
Arm/Group | Guided Arm | Non-Guided Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Screen Failures: Screen failures constitute patients who were registered to the study but were not assigned treatment for various reasons.
Arm/Group | Guided AC Sensitive | Guided TC Sensitive | Guided AC Non-sensitive | Guided TC Non-Sensitive | Non-guided AC | Non-guided TC | Screen Failures
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/7 | 3/6 | 2/6 | 1/6 | 2/7 | 1/18
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 6/6 | 6/6 | 6/6 | 7/7 | 1/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guided AC Sensitive (N=6) | Guided TC Sensitive (N=7) | Guided AC Non-sensitive (N=6) | Guided TC Non-Sensitive (N=6) | Non-guided AC (N=6) | Non-guided TC (N=7) | Screen Failures (N=18)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Ear and labyrinth disorders: ear complete hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infections and infestations: Infection with neutrophils: Abdomen NOS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infections and infestations: UTI (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 2 | 1 | 0 | 1 | 0
White blood cell decreased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guided AC Sensitive (N=6) | Guided TC Sensitive (N=7) | Guided AC Non-sensitive (N=6) | Guided TC Non-Sensitive (N=6) | Non-guided AC (N=6) | Non-guided TC (N=7) | Screen Failures (N=18)
Anemia (Blood and lymphatic system disorders) | 3 | 3 | 1 | 2 | 1 | 3 | 0
Lymph node pain (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 0
Cardiac disorders: Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac disorders: palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Blurred vision (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Dry eye (Eye disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Extraocular muscle paresis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders: eye lids twitching (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Watering eyes (Eye disorders) | 0 | 2 | 1 | 1 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0
Anal mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 5 | 4 | 3 | 4 | 3 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 4 | 1 | 3 | 1 | 3 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorders: inflamed gums (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 3 | 2 | 3 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 4 | 2 | 2 | 3 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 3 | 0 | 1 | 0 | 0
Edema face (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Edema limbs (General disorders) | 2 | 3 | 1 | 1 | 1 | 1 | 0
Edema trunk (General disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 5 | 5 | 6 | 5 | 6 | 0
Fever (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
General disorders and administration site conditions: cold intolerance (General disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 1 | 2 | 1 | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 2 | 1 | 1 | 0 | 2 | 0
Infections and infestations: UTI (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Lymph gland infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 3 | 1 | 2 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight gain (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 2 | 0 | 1 | 0 | 2 | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 5 | 1 | 5 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 2 | 0 | 4 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 1 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 2 | 0 | 5 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 1 | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder : muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 1 | 2 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 2 | 0
Dysgeusia (Nervous system disorders) | 3 | 3 | 2 | 3 | 0 | 4 | 0
Headache (Nervous system disorders) | 5 | 4 | 5 | 5 | 4 | 3 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3 | 2 | 1 | 2 | 4 | 0
Sinus pain (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 3 | 1 | 0
Depression (Psychiatric disorders) | 1 | 4 | 0 | 2 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 4 | 3 | 4 | 2 | 4 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 3 | 1 | 3 | 3 | 0 | 1
Uterine pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 6 | 3 | 3 | 3 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 2 | 1 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1 | 0 | 1 | 0
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Respiratory, thoracic and mediastinal disorders: dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 5 | 2 | 2 | 5 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 1 | 3 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 1 | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders: nose sores (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 2 | 3 | 3 | 1 | 2 | 3 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Vascular disorders: easy bruising (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular disorders: epitaxsis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes